CLINICAL TRIAL: NCT00172055
Title: Study to Assess Efficacy and Safety of Zoledronic Acid and the Value of Markers of Bone Resorption in the Prediction of Bone Metastases and Cancer Treatment-induced Bone Loss (CTIBL) in Patients With Prostate Cancer on Hormone Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446GBE03
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Cancer Prostate
Keywords: Zoledronic acid; Zometa; prostate cancer; osteoporosis
MeSH Terms: conditions — Prostatic Neoplasms; Osteoporosis | interventions — Zoledronic Acid

ARMS (1):
- ZOL446 (zoledronic acid) (Experimental)
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid

SUMMARY:
The objective of the study is to investigate whether blood markers can be used to predict the development of bone metastases and to assess the efficacy and safety of zoledronic acid in cancer treatment induced bone loss.

ELIGIBILITY:
Inclusion Criteria:

* All stages of prostate cancer without bone metastases
* No evidence of severe osteoporosis
* ECOG performance status 0, 1 or 2

Exclusion Criteria:

* Surgery / fracture at the lumbosacral spine, bilateral hip implants
* Evidence of metabolic bone diseases,
* Treatment with bisphosphonates or calcitonin within the previous year or chronic systemic corticosteroid treatment
* Abnormal kidney or liver function
* Other cancers within the last 5 years

Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2004-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
If and to what extent rising levels of the bone resorption marker CTX can be used as an indicator for the development of bone metastases, diagnosed via bone scintigraphy. | at 6 months

SECONDARY OUTCOMES:
If and to what extent rising levels of PSA can be used as an indicator for the development of bone metastases | at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (19):
- Belgium (19):
  - Novartis Investigative Site, Anderlecht
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Charleroi
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Ghent
  - Novaris Investigative Site, Gosselies
  - Novartis Investigative Site, Kortrijk
  - Novartis Investigative Site, Leper
  - Novartis Investigative Site, Leuven
  - Novaris Investigative Site, Libramont
  - Novartis Investigative Site, Mont-Godinne
  - Novartis Investigative Site, Roeselare
  - Novartis Investigative Site, Tongeren
  - Novartis Investigative Site, Tournai
  - Novartis Investigative Site, Turnhout
  - Novartis Investigative Site, Wilrijk
  - Novartis Investigative Site, Woluwe-Saint-Lambert